CLINICAL TRIAL: NCT02238535
Title: Use of Ventavis in Patients With Postembolic Residual Pulmonary Hypertension
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ventavis_PRPH
Record Dates: First submitted 2014-09-03; First posted 2014-09-12 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Residual Pulmonary Hypertension
MeSH Terms: interventions — Iloprost; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ventavis + Warfarin (Active Comparator): Patients in this group will receive drug treatment - ventavis (2,0 ml - 6 time per day - during 5 days). Warfarin - INR=2,0-3,0
  Interventions: Drug: Ventavis; Drug: Warfarin
- Warfarin (Active Comparator): Patients in this group will receive drug treatment according to up-to-date guidelines (Warfarin - INR=2,0-3,0)
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Ventavis
  Arms: Ventavis + Warfarin
Drug: Warfarin

SUMMARY:
To assess the effectiveness of the synthetic analogue of prostacyclin in postembolic residual pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pulmonary embolism after undergone surgical treatment (intravascular thrombolysis, catheter thrombus fragmentation)
* Patients with preserved thromboembolism in the pulmonary circulation system and mean pressure in the pulmonary artery of more than 25 mm Hg

Exclusion Criteria:

* Patient did not sign the informed consent.
* Mean pulmonary artery pressure after surgical treatment less than 25 mm Hg
* Age above 75 years.
* Patients with an increased risk of bleeding - including gastric ulcer and 12 duodenal ulcer in acute, hemorrhagic stroke.
* Severe coronary artery disease (unstable angina, myocardial infarction within the last 6 months).
* Acute heart failure or CHF IV in NYHA.
* Severe arrhythmias.
* Pregnancy, lactation.
* The presence of severe diseases of other organ systems that may result in death during the first year after surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-03 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Pulmonary hypertension | 6 months
  The average pressure in the pulmonary artery trunk (according to direct tensiometry before Ventavis therapy, after the therapy according to transthoracic echocardiography and six months after discharge (transthoracic echocardiography).

SECONDARY OUTCOMES:
Number of deaths | 6 months
Number of recurrent pulmonary embolisms | 6 months
Number of venous thromboembolisms | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- State Research Institute of Circulation Pathology, Novosibirsk, Russia

REFERENCES:
- See also: Related Info — http://meshalkin.ru